CLINICAL TRIAL: NCT00946829
Title: Study of Hypertensive Population Under Treatment With Micardis in Real Clinical Conditions With the Goal to Control the Early Morning BP Rise
Brief Title: Study of Hypertensive Population Under Treatment With Telmisartan in Real Clinical Conditions With the Goal to Control Early Morning Blood Pressure Rise
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 502.425
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2009-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: telmisartan

SUMMARY:
The aim of the observational study is to ascertain the degree of blood pressure control in the early-morning hours after 8 weeks of treatment with Telmisartan/Telmisartan+Hydrochlorothiazide and during 44 weeks of follow-up, in patients with hypertension using home blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate essential hypertension and whose medical condition make them eligible for treatment with Telmisartan/Telmisartan+HCTZ

Exclusion Criteria:

* Pre-menopausal women who had had no birth control, who are pregnant or nursing
* Patients with advanced hepatic impairment, advanced renal impairment or both
* Patients with functional class III or IV (NYHA) congestive heart failure (CHF), unstable angina, acute myocardial infarction, heart surgery or stroke within the previous six months
* Patients with any valvular disease with hemodynamic repercussion
* Patients receiving chronic administration of oral anticoagulants or digoxin
* Patients with known hypersensitivity to any component in the formulation of Micardis / MicardisPlus
* Patients with previous history of angioedema associated with ACE inhibitors
* Patients with severe, uncontrolled hypertension or any form of secondary hypertension
* Patients with any other clinical conditions which, in the opinion of the investigator, would not allow for the safe completion of the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 18299 (Actual)
Dates: Start 2003-01; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean early morning systolic blood pressure, mean early morning diastolic blood pressure, and degree of control. (6:00 to 11:59), BP < 135/85 mmHg. (HBPM: mean of morning measurements). | 217 Weeks

SECONDARY OUTCOMES:
Clinical control (office BP), response rates, reduction in office cuff systolic and diastolic BP. Office BP control criteria: BP < 140/90 mmHg. Pulse rate, pulse pressure, discontinuations and tolerability. | 217 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Belgium
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Canada
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Colombia
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Czechia
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Ecuador
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Indonesia
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Jordan
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Lebanon
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Mexico
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Turkey (Türkiye)
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Venezuela
- Boehringer Ingelheim Investigational Site, Boehringer Ingelheim Investigational Site, Yemen